CLINICAL TRIAL: NCT01776034
Title: Examining the Efficacy of a SystemCHANGE™ Weight Management Intervention in Stroke Survivors and Persons With Chronic Inflammatory Autoimmune/Immune-mediated Diseases
Brief Title: Health Promotion and Wellness Program for Adults With Disabling Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American Heart Association (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Matthew Plow, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-14-16 / 03-14-24
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Stroke; Multiple Sclerosis; Rheumatoid Arthritis
Keywords: Self Care; Exercise; Weight management
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SystemCHANGE Group Lifestyle counseling (Experimental): The SystemCHANGE™ intervention will be delivered over a six-month period involving 12 face-to-face group sessions (1.5 to 2 hours each) held weekly for three months, followed by three monthly "booster calls." Intervention groups include ~10 to 15 patients, and friends and family members are encouraged to attend. Intervention sessions consist of 30-min to 60-min of behavior change activities and 60-min focused on healthy behaviors.
  Interventions: Behavioral: SystemCHANGE Group Lifestyle counseling
- Phone Lifestyle Counseling (Active Comparator): Participants will receive pamphlets that contain information on healthy eating, physical activity, sleep, and symptom management, and will be followed-up with telephone calls.
  Interventions: Behavioral: Phone Lifestyle Counseling

INTERVENTIONS:
Behavioral: SystemCHANGE Group Lifestyle counseling
  Arms: SystemCHANGE Group Lifestyle counseling
Behavioral: Phone Lifestyle Counseling
  Arms: Phone Lifestyle Counseling

SUMMARY:
The objective of this study is to conduct a randomized controlled pilot study to examine the efficacy, feasibility and safety of the SystemCHANGE™(SC) health promotion and wellness program in adults with disabling conditions. Particularly, the study will focus on developing a program of research on adapting and testing SC weight management interventions in overweight and obese stroke survivors and persons with chronic inflammatory autoimmune/immune-mediated diseases, specifically those with multiple sclerosis (MS) and rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Individuals with disabling conditions, such as stroke, multiple sclerosis, or rheumatoid arthritis, face many barriers to engaging in physical activity, healthy nutritional habits, and good sleep hygiene. This leads to weight gain, de-conditioning, and declines in upper- and lower- extremity function, which makes it even more difficult to engage in healthy behaviors, thereby perpetuating a cycle of functional decline. Developing an effective weight management intervention may be a strategy for disrupting this disabling cycle and reducing the impact of the disease. Fostering a positive social environment may help adults with disabling conditions overcome barriers to engaging in healthy behaviors. SystemCHANGE (SC) is a new behavior change program that uses approaches consistent with social ecological theories and process improvement techniques (i.e. changing the dynamics of a system or group) to increase social support in lifestyle behaviors that promote energy balance. SC focuses on redesigning the social environment using a series of trial-and-error "experiments", which is in contrast to cognitive-behavioral interventions that focus on changing a person's viewpoint of a situation and increasing motivation. In a SC intervention, individuals are taught a set of skills to assist them in incorporating habitual lifestyle behaviors into their daily systems so they succeed despite wavering motivation. The rationale for developing a weight management intervention for these patients is to slow disability progression and prevent secondary conditions.

ELIGIBILITY:
Inclusion Criteria Stroke:

* Physician-confirmed diagnosis of stroke (> 6 weeks)
* Body mass index between 23 to 45 kg/m2
* Age 30 to 75 years

Exclusion Criteria Stroke:

* Pregnant or plans to become pregnant in the next 6 months
* Current participation in a face-to-face weight management program
* Uncontrolled diabetes (hospitalization within the prior 6 months)
* Serious mental illness
* Thyroid and adrenal gland diseases
* Inability to walk 3 meters with or without a cane or walker
* Severe cardiopulmonary disease that limits engagement in physical activity (e.g., myocardial infarction, congestive heart failure, coronary artery bypass grafting or valve replacement during the past three months, serious cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, and pulmonary embolus) or abnormal blood pressure or heart rate response after the 6-Minute Walking Test (e.g., a drop in systolic blood pressure of >10mmHg from baseline)
* Severe cognitive deficits (Screening questioanire called the Short Orientation Memory-Concentration < 12)
* Currently taking oral corticosteroids, antipsychotic (except for depression medication), or medications specifically for weight loss
* 3 or more falls in the past month
* Bulimia
* Unable to speak English over the phone
* Able to eat independently and is not on a special diet because of difficulty in swallowing
* Unstable weight (gained or lost >10lbs in the last two months)

Inclusion Criteria MS or RA:

* Physician-confirmed diagnosis of multiple sclerosis or rheumatoid arthritis
* Body mass index between 23 to 45 kg/m2

Exclusion Criteria MS or RA:

* Pregnant or plans to become pregnant in the next 6 months
* Current participation in a face-to-face weight management program
* Uncontrolled diabetes (hospitalization within the prior 6 months)
* Serious mental illness
* Inability to walk 3 meters with or without a cane or walker
* Severe cardiopulmonary disease that limits engagement in physical activity
* Severe cognitive deficits (Short Orientation Memory-Concentration < 12)
* Currently taking oral corticosteroids, antipsychotic (except for depression medication), or medications specifically for weight loss
* 3 or more falls in the past month
* Bulimia
* Unable to speak English
* Uncontrolled thyroid or adrenal disease (change in type and dosage of medication within the prior 3 months)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body weight. | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  A digital scale will be used to measure Body weight.

SECONDARY OUTCOMES:
Changes from baseline in cardiovascular risk biomarkers. | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  The Alere Cholestech LDX 1 Analyzer will be used to measure Triglycerides levels.
Changes from baseline in Walking Test. | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  A Six Minute Walking Test will be administered using standardized instructions and verbal cues
Changes from baseline in 1-minute sit to stand test | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  A 1-minute sit to stand test will be administered using standardized instructions and verbal cues
Changes from baseline Physical Activity | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  Physical Activity and Disability Survey-Revised will be administered to assess physical function. Higher scores on the Physical Activity and Disability Survey-Revised indicates increased physical activity levels. Score range: Not applicable.
Changes from baseline Self-efficacy for weight management | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  Weight Efficacy Lifestyle Questionnaire-Short Form (WEL-SF) will be administered. A higher score on the weight efficacy lifestyle questionnaire indicates more confidence to engage in a healthy behavior (possible score range for self-efficacy weight is 1 to 10)
Changes from baseline social support for physical activity from family | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  Social Support for Exercise Behavior scales will be administered. A higher score on social support scales indicates greater social support from family to engage in physical activity (possible score range is 1 to 5).
Changes from baseline in emotional well-being | Each patient will be given the assessments at 2 points during the study, at baseline and at posttest (an average of 6 months from baseline).
  Quality of Life in Neurological Disorders (Neuro-Qol) positive affect & wellbeing questionnaires will be administered. Higher scores on Quality of Life in Neurological Disorders (Neuro-Qol) positive affect and well-being indicates a greater life satisfaction (possible score range 9 to 45).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Plow, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plow M, Moore SM, Kirwan JP, Frost F, Katzan I, Jaeger S, Alberts J. Randomized controlled pilot study of a SystemCHANGE weight management intervention in stroke survivors: rationale and protocol. Trials. 2013 May 7;14:130. doi: 10.1186/1745-6215-14-130. PMID 23782741